CLINICAL TRIAL: NCT01991314
Title: Treatment of Iron Deficiency Anaemia in Adults and Adolescents With Inflammatory Bowel Disease Using Ferrous Sulphate: Tolerance and Effects on Haemoglobin, Mood, Quality of Life and Fatigue
Brief Title: Treatment of Iron Deficiency Anaemia in Inflammatory Bowel Disease With Ferrous Sulphate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-023797-39
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2015-11

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — ferrous sulfate

STUDY DESIGN:
Masking Description: This was an open label trial
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferrous sulphate (Experimental): Ferrous sulphate 200mg twice daily for 6 weeks
  Interventions: Drug: Ferrous sulphate

INTERVENTIONS:
Drug: Ferrous sulphate — 200mg tablets.

SUMMARY:
Iron deficiency anaemia is common in inflammatory bowel disease (IBD), affecting at least 20% patients at any one time. Hepcidin, a recently described anti-microbial peptide synthesized by the liver, is a key regulator of iron homeostasis. It interferes with absorption of iron into enterocytes, macrophages and hepatocytes by binding to ferroportin. Hepcidin levels rise when total body iron levels rise and protect against iron overload; conversely, in iron deficiency, levels are low. Hepcidin levels also rise under the influence of interleukins (IL)-6 and -1, a factor likely to contribute to iron deficient erythropoesis in active IBD. Whether hepcidin levels predict resistance to oral iron therapy in IBD is unknown, though it may impair its immediate oral absorption. Adult IBD patients who are anaemic report quality of life and fatigue scores comparable to those seen in malignancy.

IBD diagnosed in adolescence interferes with growth, education and employment as well as psychosocial and sexual development. Not surprisingly, adolescents with IBD have a high prevalence of psychological distress, particular depression. Limited historical, and our own data suggest that children and adolescents with IBD are more anaemic than adults, and less often treated with oral iron. What is not clear is whether the apparent under-utilisation of oral iron in paediatric care is because of a perceived lack of benefit or doctors' concerns about possible side effects including worsening disease activity.

To address these questions, the investigators propose a comparative study of 6 weeks of oral iron supplementation in adolescents and adults with iron deficiency anaemia in IBD. Patients will be given oral iron supplementation. Before and after iron therapy, the investigators shall assess haemoglobin concentrations; IBD activity; quality of life (QOL), perceived stress, mood and fatigue; iron metabolism, including serum hepcidin.

DETAILED DESCRIPTION:
Methods Before and after iron therapy, we assessed haemoglobin concentrations; iron status markers; serum hepcidin concentration; IBD activity; iron tolerance; and QOL, perceived stress, mood, coping and fatigue using psychometric questionnaires.

Patients. Patients aged 13 - 18 years were defined as adolescents, and those aged ≥ 19 years as adults. Between January 2012 and April 2015, patients with IBD (ulcerative colitis (UC), Crohn's disease or IBDU (IBD unclassified) diagnosed by standard clinical, radiological and pathological criteria) who within the next month were due to attend the adult, young people's and paediatric IBD clinics at Barts and the Royal London Hospitals, Barts Health Trust or the paediatric IBD clinic at Chelsea and Westminster NHS Trust, London, UK, were screened for the result of their haemoglobin concentration at their previous clinic attendance. Those found to be anaemic were sent a letter of explanation about, and invitation to participate in, the trial. They were telephoned 1-2 weeks after this letter was sent to them and asked about current and previous iron therapy: those apparently eligible (see below) and verbally consenting to participate were then seen by a trial doctor or research nurse either at their next clinic appointment, or on another mutually convenient occasion. Informed written consent from the patients or their parents, as appropriate, was obtained at this meeting, and patients who remained eligible on the basis of their iron therapy history and clinical, and haematological criteria were enrolled in the trial.

Definition of iron deficiency anaemia: Anaemia was defined by age and sex-adjusted World Health Organisation criteria (males <13.0 g/dl; females and children aged 13 years <12.0 g/dl) (WHO 2001). For inclusion in the trial, patients had to be both anaemic and have transferrin saturation <18%. They also had to report either tolerance of previous course(s) of oral iron, or to be naïve to this treatment.

Exclusion criteria: Patients were excluded if they did not meet the haematological inclusion criteria on the admission-to-study blood test ('screening failures'), if they had been given oral or intravenous iron within 3 months, or if they had previously been intolerant of oral iron. Other exclusion criteria were age <13 years, vitamin B12 or folate deficiency, anaemia caused by drugs used to treat IBD, haemoglobinopathy, presence of stoma or ileoanal pouch, severely active IBD requiring hospital admission from clinic, severe cardiopulmonary, hepatic, renal or other disease, pregnancy, breast-feeding, use of cholestyramine, and inability to speak English well enough to complete the consent form or psychometric questionnaires.

Regulatory and funding considerations: The trial was approved by the Southampton National Research Ethics Committee (number 10/H504/90 and EUDRACT number 2010-023797-39) and was necessarily registered as a Clinical Trial of an Investigational Medical Product (CTIMP) with the Medicines and Healthcare Products Regulatory Agency (number 14620/0035/001-0001) and ClinTrials.Gov. The trial was sponsored by Barts Health NHS Trust. The trial was kindly funded by a grant from Core and British Society for Paediatric Gastroenterology, Hepatology and Nutrition.

Trial protocol and treatment. At enrolment, demographic data including age, sex, disease type, education, marital status, smoking habit, weight and height were recorded. Disease type, location, behaviour and extent, using Montreal classifications (Silverberg 2005) and previous surgeries were noted from medical records. Patients completed six psychometric questionnaires to assess mood, fatigue and quality of life (QOL): the Hospital Anxiety and Depression Scale (HADS-A and HADS-D)(Zigmond 1983, Bjelland 2002), the recent and general Perceived Stress Questionnaires (PSQ-R and PSQ-G) (Levenstein 1993), the Patient Health Questionnaire (PHQ-9) (Kroenke 2001), the Coping Inventory for Stressful Situations (CISS)(Endler 2000), the Big Five Inventory (BFI) (Ramstedt or one of the John refs - check which is right), the Multi-dimension Fatigue Inventory (MFI) (Smets 1995) and the Short Inflammatory Bowel Disease Questionnaire (SIBDQ)(Irvine 1996). Symptomatic disease activity was assessed using the Harvey-Bradshaw Index (HBI) for patients with Crohn's disease (Harvey 1998), and Simple Clinical Colitis Activity Index (SCCAI) for those with ulcerative colitis (Walmsley 2001). Blood was collected for blood count, including haemoglobin, iron studies and hepcidin, and C-reactive protein (CRP); and a stool sample was obtained for faecal calprotectin, as an objective measure of disease activity (Kopylov 2014). Patients were given 6 weeks treatment with 200mg oral ferrous sulphate (Wockhardt Ltd, Ranbaxy Ireland Ltd) twice daily.

After one week, patients were telephoned to assess tolerance to treatment: those intolerant of or non-adherent to oral iron were withdrawn from the trial and asked to attend for repeat blood tests, questionnaires and faecal calprotectin as end of trial measures. After 6 weeks of iron treatment, the above measurements were repeated and adherence assessed by counting of returned iron tablets.

Outcome measures. The primary outcome measure was mean increase in haemoglobin concentration in the adolescent and adult groups after 6 weeks of treatment. Secondary outcome measures in the two groups were tolerance of oral iron; changes in disease activity (HBI, SCCAI, CRP, faecal calprotectin), SIBDQ, HADS-A, HADS-D, PSQ-R, PSQ-G, PHQ-9, CISS, BFI and MFI scores, and relation of serum hepcidin at baseline to haemoglobin response to oral iron. The SCCAI was used for scoring clinical disease activity in the three adolescent patients with IBDU.

Assays Haemoglobin, iron studies and routine biochemistry were measured in the haematology and biochemistry laboratories at the Royal London and Chelsea and Westminster Hospitals. Serum for hepcidin assays was stored at -800 C until assay in duplicate in the University Birmingham by mass spectrometry (Ward 2008). The mass spectrometer was calibrated at each assay but because it is not serviced annually, the Research & Development Department at Barts Health NHS Trust insists on the statement herein that the hepcidin assay did not meet strict GCP compliance regulations. Stool samples were stored at -800 C until the end of recruitment: they were then extracted and quantified for calprotectin in duplicate by ELISA (ACCUSAY Calprotectin, Launch Diagnostics, Ltd, Longfield, UK) in the Clinical Immunology laboratory at Royal London Hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients with proven iron deficiency anaemia on World Health Organisation (WHO)criteria Patients aged 13 - 18 will be considered adolescents, and aged >18 as adults.

Exclusion Criteria:

Anaemia caused by B12 or folate deficiency, or secondary to drugs used to treat IBD; haemoglobinopathies or myelodysplasia; severe cardiopulmonary, hepatic or renal disease; severe cardiopulmonary, hepatic or renal disease; pregnancy and breast feeding females.

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Rampton, DPhil, FRCP, Principal Investigator — Queen Mary London
Locations (1):
- Barts Health NHS Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rampton DS, Goodhand JR, Joshi NM, Karim AB, Koodun Y, Barakat FM, Macken L, Ward DG, Iqbal TH, Epstein J, Fell JM, Sanderson IR. Oral Iron Treatment Response and Predictors in Anaemic Adolescents and Adults with IBD: A Prospective Controlled Open-Label Trial. J Crohns Colitis. 2017 Jun 1;11(6):706-715. doi: 10.1093/ecco-jcc/jjw208. PMID 27932449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2012 and April 2015; adult and paediatric IBD clinics at Barts and the Royal London Hospitals, or the paediatric IBD clinic at Chelsea and Westminster NHS Trust, London, UK, w
Pre-assignment Details: After trial closure, 1 adult (transferrin saturation 22%) and 1 adolescent (Hb 12.0) were found to have been recruited in error and were excluded from further analysis, leaving 88 participants in total.
Groups:
- Adolescents - Ferrous Sulphate: 45 adolescents (13-18 years) given ferrous sulphate 200mg bd for 6 weeks
- Adults - Ferrous Sulphate: 43 adults (>18 years) given ferrous sulphate 200mg bd for 6 weeks
Period: Overall Study
Arm/Group | Adolescents - Ferrous Sulphate | Adults - Ferrous Sulphate
Started | 45 | 43
Completed | 34 | 32
Not Completed | 11 | 11
Not completed — Adverse Event | 5 | 1
Not completed — Lost to Follow-up | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Adolescent - Ferrous Sulphate: 45 adolescents (age 13-18 years) given oral ferrous sulphate 200mg bd for 6 weeks
- Adults - Ferrous Sulphate: 43 adults (age >18 years) given oral ferrous sulphate 200mg bd for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Adolescent - Ferrous Sulphate | Adults - Ferrous Sulphate | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45 | 0 | 45
  Between 18 and 65 years | 0 | 40 | 40
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 23 | 20 | 43
Region of Enrollment [Number; unit: participants]
  United Kingdom | 45 | 43 | 88

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Haemoglobin Concentration.
Description: Change in serum Hb concentration in g/dl after 6 weeks of oral iron
Time Frame: Baseline (0 weeks) and end of trial (6 weeks)
Population: Intention to treat population
Measure: Mean (Standard Error); unit: g/dl
Groups:
- Adolescents: Patients aged 13 - 18 years
- Adults: IBD patients aged >18
Arm/Group | Adolescents | Adults
Number analyzed (Participants) | 45 | 43
g/dl | 1.22 (0.21) | 1.30 (0.27)
Statistical Analysis 1: Comparison: Adolescents vs Adults; Test type: Non-Inferiority or Equivalence — We calculated, on the premise that there is non-inferiority between adolescent and adult groups in the difference in increase of mean haemoglobin levels of 0.35g/dL, with estimated standard deviation 0.7g/dL following treatment, that 45 patients in each group would be required, derived using power 80% power, 1-sided significance level 0.05 and R 0.5 for the covariate; this calculation took into account planned ANCOVA methodology and 20% patients who might be lost to follow up or withdraw; p = 0.23, ANCOVA — To test the hypothesis of non-inferiority with maximal statistical power, ANCOVA (one-tailed P<0.05) was employed to compare the change in mean haemoglobin levels between adults and adolescents after accounting for necessary covariates; Mean Difference (Net) = 0.08

2. Secondary Outcome: Intolerance of Oral Iron
Description: Numbers of patients who reported intolerance of oral iron (abdominal pain, nausea, vomiting, constipation, diarrhoea or headache)
Time Frame: Baseline (0 weeks) to end of trial (6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Adolescents | Adults
Number analyzed (Participants) | 45 | 43
Participants | 10 | 8
Statistical Analysis 1: Comparison: Adolescents vs Adults; Chi squared test or Fisher's exact test, as appropriate; Test type: Superiority or Other; p < 0.05, Fisher Exact; Fisher's exact test was used to compare proportions (expressed as percentages) of total number of participants in each group who were iron intolerant; difference in proportions = 3.6

3. Secondary Outcome: Change in Disease Activity (Stool Calprotectin)
Description: Difference between faecal calprotectin measured at baseline and at end of study
Time Frame: Baseline (0 weeks) and end of trial (6 weeks)
Population: Per protocol analysis
Measure: Mean (Standard Error); unit: ug/g
Arm/Group | Adolescents | Adults
Number analyzed (Participants) | 34 | 32
ug/g | -35 (38) | -40 (81)
Statistical Analysis 1: Comparison: Adolescents vs Adults; Unpaired Students t test; Test type: Superiority or Other; p = 0.96, t-test, 2 sided; Mean Difference (Net) = -5

4. Secondary Outcome: Change in Quality of Life Score
Description: Short Inflammatory Bowel Disease Questionnaire (SIBDQ score), a health-related quality of life tool measuring physical, social, and emotional status (summated to produce a score of minimum 10 to maximum 70, representing poor to good quality of life, respectively). (Reporting of individual domain subscores is not valid).
Time Frame: Baseline (0 weeks) to end (6 weeks)
Population: Per protocol analysis
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Adolescents | Adults
Number analyzed (Participants) | 34 | 32
scores on a scale | 3.2 (2.6) | 5.7 (2.0)
Statistical Analysis 1: Comparison: Adolescents vs Adults; Mann-Whitney U test; Test type: Superiority or Other; p = 0.49, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 2.5

5. Secondary Outcome: Changes in Anxiety
Description: Hospital Anxiety and Depression Score (HADS)-A, a scale of 7 questions score 0-3 each, so that total score 0 is good and 21 very severe anxiety.
Time Frame: Baseline (0 weeks) and end of trial (6 weeks)
Population: Per protocol
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Adolescents | Adults
Number analyzed (Participants) | 34 | 32
units on a scale | -0.7 (0.5) | -1.1 (0.7)
Statistical Analysis 1: Comparison: Adolescents vs Adults; Mann Whitney U test; Test type: Superiority or Other; p = 0.85, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.4

6. Secondary Outcome: Changes in Fatigue
Description: Multidimensional Fatigue Inventory (MFI) is a 20 question-based scale with total scores ranging between 20 (very good) and 100 (very severe fatigue).
Time Frame: Baseline (0 weeks) and end of trial (6 weeks)
Population: Per protocol
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Adolescents | Adults
Number analyzed (Participants) | 34 | 32
units on a scale | 0.9 (1.4) | 1.9 (0.7)
Statistical Analysis 1: Comparison: Adolescents vs Adults; Mann Whitney U test; Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -1.0

7. Secondary Outcome: Changes in Stress Levels
Description: Perceived Stress Questionnaire (PSQ)-G is a 30-question measure of perceived stress giving total scores ranging between 30 (very unstressed) to 120 (very stressed).
Time Frame: Baseline (0 weeks) and end of trial (6 weeks)
Population: Per protocol analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Adolescents | Adults
Number analyzed (Participants) | 34 | 32
units on a scale | 4.1 (2.5) | -11.8 (2.5)
Statistical Analysis 1: Comparison: Adolescents vs Adults; Mann-Whitney U test; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -15.9

ADVERSE EVENTS:
Time Frame: Baseline (0 weeks) to end of trial (6 weeks)
Description: Patients were asked to contact us by telephone if they had symptoms suggesting adverse events (eg abdominal pain, nausea, vomiting, constipation, diarrhea, headache), or if their Crohn's disease or ulcerative colitis symptoms were worsening. Patients described their own symptoms and were not prompted by a checklist or other systematic questionnaire.
Arm/Group | Adolescents | Adults
Serious Adverse Events (participants affected / at risk) | 2/45 | 1/43
Other Adverse Events (participants affected / at risk) | 8/45 | 7/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents (N=45) | Adults (N=43)
Crohn's patient admitted to hospital with abdominal pain and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's patient admitted to hospital with abdominal pain, vomiting and constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcerative colitis patient admitted with flare of her colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescents (N=45) | Adults (N=43)
AE (Gastrointestinal disorders) | 8 (8) | 7 (7) — Crohn's or UC patients with abdominal pain (n=8), constipation (n=3), diarrhoea (n=4), nausea (n=2), vomiting (n=1) and/or headache (n=1). [Note that several patients had more than 1 AE symptom].

LIMITATIONS AND CAVEATS:
Findings may not be generalizable. Trial not blinded. We studied patients who had tolerated oral iron before or were naïve to it. Only half of patients returned tablet containers for counting. Questionnaires used not validated for young people.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes